CLINICAL TRIAL: NCT04079530
Title: A Multicenter, Randomized, Active-controlled, Single-blind, 2-Period, 12-Sequence Crossover Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Pemafibrate in Patients With Dyslipidemia
Brief Title: A Clinical Pharmacology Study of K-877 Controlled Release Tablet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: K-877-CR-01
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Treatment A (Experimental): Period1:K-877 IR 0.2 mg/day, Period2:K-877 CR 0.4 mg/day (pre-meal)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.4 mg/day
- Treatment B (Experimental): Period1:K-877 IR 0.2 mg/day, Period2:K-877 CR 0.4 mg/day (postprandial)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.4 mg/day
- Treatment C (Experimental): Period1:K-877 IR 0.2 mg/day, Period2:K-877 CR 0.8 mg/day (pre-meal)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment D (Experimental): Period1:K-877 IR 0.2 mg/day, Period2:K-877 CR 0.8 mg/day (postprandial)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment E (Experimental): Period1:K-877 CR 0.4 mg/day, Period2:K-877 IR 0.2 mg/day (pre-meal)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.4 mg/day
- Treatment F (Experimental): Period1:K-877 CR 0.4 mg/day, Period2:K-877 IR 0.2 mg/day (postprandial)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.4 mg/day
- Treatment G (Experimental): Period1:K-877 CR 0.4 mg/day, Period2:K-877 CR 0.8 mg/day (pre-meal)
  Interventions: Drug: K-877 CR 0.4 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment H (Experimental): Period1:K-877 CR 0.4 mg/day, Period2:K-877 CR 0.8 mg/day (postprandial)
  Interventions: Drug: K-877 CR 0.4 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment I (Experimental): Period1:K-877 CR 0.8 mg/day, Period2:K-877 IR 0.2 mg/day (pre-meal)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment J (Experimental): Period1:K-877 CR 0.8 mg/day, Period2:K-877 IR 0.2 mg/day (postprandial)
  Interventions: Drug: K-877 IR 0.2 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment K (Experimental): Period1:K-877 CR 0.8 mg/day, Period2:K-877 CR 0.4 mg/day (pre-meal)
  Interventions: Drug: K-877 CR 0.4 mg/day; Drug: K-877 CR 0.8 mg/day
- Treatment L (Experimental): Period1:K-877 CR 0.8 mg/day, Period2:K-877 CR 0.4 mg/day (postprandial)
  Interventions: Drug: K-877 CR 0.4 mg/day; Drug: K-877 CR 0.8 mg/day

INTERVENTIONS:
Drug: K-877 IR 0.2 mg/day — K-877 IR 0.1 mg tablet
  Other Names: Pemafibrate
  Arms: Treatment A; Treatment B; Treatment C; Treatment D; Treatment E; Treatment F; Treatment I; Treatment J
Drug: K-877 CR 0.4 mg/day — K-877 CR 0.4 mg tablet
  Other Names: Pemafibrate
  Arms: Treatment A; Treatment B; Treatment E; Treatment F; Treatment G; Treatment H; Treatment K; Treatment L
Drug: K-877 CR 0.8 mg/day — Two K-877 CR 0.4 mg tablet
  Other Names: Pemafibrate
  Arms: Treatment C; Treatment D; Treatment G; Treatment H; Treatment I; Treatment J; Treatment K; Treatment L

SUMMARY:
A study to compare the efficacy, safety, and pharmacokinetics of K-877 controlled release tablets with a current normal K-877 tablet in dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dyslipidemia had to be age 20 years or older at written informed consent(ICF)
2. Men and postmenopausal women.
3. Patients who have received dietary or exercise guidance from 12 weeks prior to Screening.
4. Patients who have clinical laboratory records with fasting serum TG ≥ 150 mg / dL (or ≥ 200 mg / dL if not fasting) within 6 months before written informed consent.
5. Patients with a fasting serum TG ≥ 150 mg / dL at Screening.

Exclusion Criteria:

1. Patients with a fasting serum TG ≥ 500 mg / dL at Screening
2. Patients who require administration of prohibited drugs during the clinical trial period after written informed consent
3. Patients who have malabsorption or those who have had the history, or who have undergone other surgical procedures that may affect absorption (excluding appendectomy or hernia treatment etc)
4. Patients with uncontrolled thyroid disease
5. Patients with uncontrolled diabetes as defined by a HbA1c(NGSP) ≥ 8.0％ at Screening
6. Persons with uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg)
7. Patients with an AST or ALT three times the upper limit at Screening
8. Patients with cirrhosis or those with biliary obstruction
9. Patients with malignant tumor or those who are judged to have a high risk of recurrence
10. Patients who have collected 400 mL or more of whole blood within 16 weeks, or 200 mL or more of whole blood within 4 weeks, or blood samples (plasma and platelet components) within 2 weeks before Screening
11. Patients with a history of serious drug allergies (anaphylactic shock, etc.)
12. Patients with a history of hypersensitivity to pemafibrate, patients who have stopped taking pemafibrate for reasons of insufficient efficacy or safety
13. Patients who participate in other clinical trials at the time of written informed consent or who have received clinical trials other than placebo for less than 16 weeks
14. Patients who have been determined inappropriate by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Efficacy: % change from baseline in fasting serum TG(mg/dL) | 4 week after administration in each period

SECONDARY OUTCOMES:
% change from baseline in fasting HDL-C levels(mg/dL) | 4 week after administration in each period
% change from baseline in fasting LDL-C levels(mg/dL) | 4 week after administration in each period
% change from baseline in fasting non-HDL-C levels(mg/dL) | 4 week after administration in each period
% change from baseline in fasting Total Cholesterol levels(mg/dL) | 4 week after administration in each period

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Japan

REFERENCES:
- [Result] Yamashita S, Araki E, Arai H, Yokote K, Tanigawa R, Saito A, Suganami H, Minamikawa S, Ishibashi S. Clinical Pharmacology of Pemafibrate Extended-release Formulation in Patients with Hypertriglyceridemia-A Phase 2, Multicenter, Active-controlled, Randomized, Single-blind, Crossover study. J Atheroscler Thromb. 2025 Mar 1;32(3):367-384. doi: 10.5551/jat.65001. Epub 2024 Sep 26. PMID 39322570